CLINICAL TRIAL: NCT06779682
Title: Feasibility Study: Systematic Screening for Obstructive Sleep Apnea (OSA) During Preoperative Consultation
Brief Title: Systematic Screening for Obstructive Sleep Apnea During Preoperative Consultation Using AI-preoperative Agents
Acronym: DASCA
Status: Active, not recruiting | Type: Observational
Sponsor: Intelligence Anesthesia (Industry)
Collaborators: Department of Anesthesiology, Hopital Foch, Suresnes, France. (Unknown); GCS Ramsay Santé pour l'Enseignement et la Recherche (Other); Hôpital privé Claude Galien - Quincy-sous-Sénart (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-A01959-30
Record Dates: First submitted 2025-01-13; First posted 2025-01-16 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Obstructive Sleep Apnea; Preoperative Evaluation
Keywords: preoperative; STOP-BANG score; Obstructive Sleep Apnea; AI; OSA
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to evaluate the feasibility of a systematic screening protocol for Obstructive Sleep Apnea (OSA) during preoperative anesthesia consultations in adults aged 50 and older undergoing elective surgery. The main questions it aims to answer are:

* Does the systematic screening protocol increase the proportion of patients identified as being at high risk for OSA compared to standard care?
* What is the impact of systematic screening on postoperative outcomes, including complications, length of stay, and mortality?

Researchers will compare standard care practices (before implementation) to the systematic screening protocol (after implementation) to determine the effect on OSA detection rates and clinical outcomes.

Participants will:

* Complete the STOP-BANG questionnaire during their anesthesia consultation.
* (Optional) Have a facial photograph taken to analyze morphometric characteristics that may correlate with OSA risk.
* Be referred for further diagnostic testing if identified as high-risk for OSA.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a national health identifier affiliated with the social security system, aged over 18, including French individuals over 50 years old, in scheduled anesthesia consultation with STOP BANG > 5 or > 4 with BMI > 35

Exclusion Criteria:

* Refusal to participate in the study, age under 50, not affiliated with the social security system, minor or under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a STOP BANG > 5 or > 4 associated with an obesity (BMI > 35 kg/m2)
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
proportion of participants in whom the risk of OSA (Obstructive Sleep Apnea Syndrome) was detected in the control group before versus the group after | From enrollment to the end of treatment at 7 months

SECONDARY OUTCOMES:
Mortality at 3 months. | From enrollment to the end of treatment at 7 months
Postoperative length of stay. | From enrollment to the end of treatment at 7 months
Sensitivity, specificity, and concordance rate of OSA (Obstructive Sleep Apnea Syndrome) detection. | From enrollment to the end of treatment at 7 months
Correlation between facial morphotype and OSA diagnosis with and without facial morphotype measurement. | From enrollment to the end of treatment at 7 months
Postoperative complications and mortality at 3 months. | From enrollment to the end of treatment at 7 months
Postoperative complications | From enrollment to the end of treatment at 7 months
  Pulmonary event Cardiac event Kidney event Vascular event

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Privé Claude Galien, Quincy-sous-Sénart, France